CLINICAL TRIAL: NCT02773121
Title: Feasibility of Using Physical Activity Monitoring for Enhancing Cognition in Healthy Seniors
Brief Title: Physical Activity and Cognition Study
Acronym: CTSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-34352
Record Dates: First submitted 2016-05-11; First posted 2016-05-16 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Aging
Keywords: Cognition; Learning; Memory; Executive Function; Attention; Neuropsychological Tests; Physical Activity; Physical Fitness; Exercise; Resistance Training; Walking; Muscle Stretching Exercises; Exercise Test; Balance; Flexibility; Body Composition
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity monitoring (Experimental): Participants will wear a physical activity sensor on the hip or waist with a belt. They will be instructed to increase their physical activity level to at least 150 min of moderate-intensity physical activity per week. They will be asked to follow guidelines in the "Go4Life" brochure, website, and/or videos by the National Institute on Aging. Participants will receive weekly phone calls to monitor their progress, to provide feedback, and to suggest example exercises.
  Interventions: Behavioral: Physical Activity
- Flexibility and balance (Active Comparator): Participants will wear a physical activity sensor on the hip or waist with a belt. They will be instructed to increase their balance and flexibility over the 12 week period of the intervention. They will be asked to follow guidelines in the "Go4Life" brochure, website, and/or videos by the National Institute on Aging. Participants will receive weekly phone calls to monitor their progress, to provide feedback, and to suggest example exercises.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Trainer-guided at-home behavioral intervention

SUMMARY:
The goal of this research study is to examine whether an intervention to increase physical activity using a body-worn sensor affects cognitive (thinking) processes.

DETAILED DESCRIPTION:
The overall duration of participation in this research study is approximately 4 months. During this time, three study visits will be required. The first visit is for informed consent and screening, the second visit is for baseline fitness and cognitive testing, and the third visit is for follow-up fitness and cognitive testing after a 12-week physical activity monitoring program. Participants will be randomized to one of two study arms, a physical activity monitoring arm and a flexibility and balance arm. Both study arms involve wearing a physical activity sensor and monitoring physical activity for a duration of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Age between 55-85 years
* Sedentary status (physically inactive; not participating in at least 30 minutes of moderate intensity physical activity on at least three days per week for at least three months)
* Generally healthy men and women
* Living in the greater Boston area
* Available for the 4 month duration of the study
* Native-English speaking or fluent in English (must have attended elementary school and higher in English)

Exclusion Criteria:

* Poor vision that cannot be corrected with glasses or contact lenses
* Presence of an acute infection
* Diagnosis of kidney failure
* Diagnosis of liver disease
* Diagnosis of thyrotoxicosis/hyperthyroidism
* Diagnosis of cancer
* Past or present conditions that affect cognitive functioning:

  1. learning disability
  2. neurological disorders or conditions (movement disorder, history of head trauma or stroke, epilepsy, etc.)
  3. psychiatric disorders or conditions (depression, anxiety disorder, etc.)
* Past or present conditions that are counter indicators for participation in cardio-respiratory fitness assessment and moderate-intensity physical activity:

  1. heart conditions (e.g. heart attack, arrhythmias, etc.)
  2. circulatory conditions (e.g. uncontrolled hypertension, leg claudication, high cholesterol, etc.)
  3. respiratory conditions (e.g., asthma or lung conditions, such as chronic obstructive pulmonary disease, acute bronchitis, acute common cold, lung cancer, pneumonia, etc.)
  4. current musculoskeletal impairments (e.g. fractures, hemiplegia, chronic joint pain, arthritis, osteoporosis, not able to walk comfortably without assistance, etc.)
  5. diagnosis of electrolyte disorder or abnormality
  6. presence of diabetes mellitus
* Obesity
* Prescription medication or other drugs that treat heart, lung, or circulatory conditions (e.g. beta blockers, bronchodilators, etc.)
* Prescription medication or other drugs that affect chemicals in the brain (e.g. antidepressants, anxiolytics, etc.)
* Implanted medical devices, such as a pacemaker or defibrillator
* Unavailable for the approx. 4-month duration of the study

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Cognition | 80-90 minutes
  Change in cognitive task performance post-intervention compared to baseline
Aerobic Fitness | 30 minutes
  Change aerobic fitness measured with treadmill test post-intervention

SECONDARY OUTCOMES:
Functional fitness: Five Times Sit to Stand | 10 min
  Change in performance in the Five Times Sit to Stand test post-intervention
Functional fitness: Timed Get Up and Go | 10 min
  Change in performance in the Timed Get Up and Go test post-intervention compared to baseline
Functional fitness: Flexibility | 10 min
  Change in performance in the Sit and Reach test post-intervention
Physical activity | 12 weeks
  Greater overall moderate-intensity physical activity time and step count and lower sedentary time in the physical activity monitoring than the flexibility and balance group

OTHER OUTCOMES:
Gait: step and stride time | 12 weeks
  Change in step and stride time over 12 weeks
Gait: stride time variability | 12 weeks
  Change in stride time variability over 12 weeks
Gait: gait symmetry | 12 weeks
  Change in gait symmetry over 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karin Schon, Ph.D., Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kern KL, Storer TW, Schon K. Cardiorespiratory fitness, hippocampal subfield volumes, and mnemonic discrimination task performance in aging. Hum Brain Mapp. 2021 Mar;42(4):871-892. doi: 10.1002/hbm.25259. Epub 2020 Dec 16. PMID 33325614
- See also: Brain Plasticity and Neuroimaging Laboratory at Boston University — http://sites.bu.edu/brainplasticity/contact-us/